CLINICAL TRIAL: NCT04721171
Title: Effectiveness of Electrical Neurostimulation as an Opioid-Sparing Alternative in the Treatment of Cyclic Vomiting Syndrome.
Brief Title: Effectiveness of Electrical Neurostimulation in Cyclic Vomiting Syndrome.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted prematurely Due to COVID-19 and Investigator left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Thangam Venkatesan, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00032752
Record Dates: First submitted 2019-04-23; First posted 2021-01-22 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Cyclic Vomiting Syndrome
MeSH Terms: conditions — Familial cyclic vomiting syndrome

STUDY DESIGN:
Intervention Model Description: Sham versus real device
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Intervention group (Active Comparator): The Bridge device is a non-invasive percutaneous electrical nerve field stimulation (PENFS) applied to the external ear. The Bridge device delivers low voltage (3.2), continuous stimulation for 5 days (around the clock) in alternating frequencies (1-10Hz) with an impulse interval of 100ms/2 sec. This is placed on the ear as per standard protocol at the beginning of the study and removed by the patient after 5 days.
  Interventions: Device: The Bridge device
- Placebo Group (Sham Comparator): The sham is similar in appearance to the Bridge device but does not deliver any electrical stimulation and is a sham that is designed to look identical to the Bridge device. It is placed on the external ear at the beginning of the study and removed by the patient after 5 days.
  Interventions: Device: The Bridge device

INTERVENTIONS:
Device: The Bridge device — he Bridge device is a non-invasive percutaneous electrical nerve field stimulation (PENFS) applied to the external ear. The Bridge device delivers low voltage (3.2), continuous stimulation for 5 days (around the clock) in alternating frequencies (1-10Hz) with an impulse interval of 100ms/2 sec. This is placed on the ear as per standard protocol at the beginning of the study and removed by the patient after 5 days.

SUMMARY:
We hypothesize that 1) Neurostimulation via a novel auricular percutaneous electrical nerve field stimulation (PENFS) device is a safe, non-invasive opioid-sparing alternative therapy for severe abdominal pain, nausea, and vomiting associated with CVS and will reduce the need for opioids. We also hypothesize that 2) PENFS reduces the length of stay (LOS), and improves patient satisfaction. We propose the following specific aim:

Aim 1. Investigate the efficacy of PENFS compared to a sham in patients with CVS seen in the ED or in the clinic or hospitalized with an acute CVS episode.

Objectives:

1. Demonstrate reduction in abdominal pain, nausea, and vomiting using validated tools.
2. Obviate or reduce the need for opioids.
3. Reduce the length of hospital stay and improve patient satisfaction.

This approach will specifically address the current opioid problem using a novel, non-invasive neurostimulation therapy with proven efficacy for opioid withdrawal. Long-term, it may improve health care outcomes and significantly reduce overall health care costs.

DETAILED DESCRIPTION:
Opioid use in CVS and the critical need for opioid sparing therapy

Given the lack of knowledge about pathophysiology and evidence-based therapies, patients are often hospitalized to treat symptoms of CVS. During an episode, patients present with severe vomiting and abdominal pain and are treated empirically with IV fluids, antiemetics, benzodiazepines, and opioids. Estimates of opioid use range from 23%-27% in adults with CVS. Patients are often dissatisfied with the level of analgesia as recurrent opioid use results in tolerance and dependence. This often undermines the physician-patient relationship and patients even leave against medical advice out of frustration with what they perceive as ineffective care. This can lead to worse outcomes including recurrent hospitalizations, morbidity and increased health care costs.

Preliminary data from a study by our group reveals that of 101 patients hospitalized with CVS at Froedtert Hospital, chronic opioid therapy is associated with a two-fold increased risk of hospitalization (RR 2.22, CI 1.1-4.4, P=0.02) and three-fold increase in hospital length of stay (LOS) (RR 3.43, CI 1.26-9.34, P=0.01). In a study of 132 CVS patients, opioid use was associated with non-response to amitriptyline (53% vs 15%, p<0.05), a prophylactic therapy used in CVS. This in turn was associated with increased frequency and duration of CVS episodes per year and increased number of hospitalizations/emergency department (ED) visits at baseline (18% vs 15.2%, p<0.05). Hence there is an urgent need for an opioid-sparing, non-invasive strategy to treat CVS symptoms.

In summary, CVS is common and disabling and is associated with significant health care costs. Our proposed project using a novel, non-invasive device to treat CVS will also address the current opioid crisis.

ELIGIBILITY:
Inclusion Criteria

• Patients who meet Rome criteria for cyclic vomiting syndrome and are in an acute episode.

Exclusion Criteria:

* Developmental delay
* Non-English speaking patients
* Pregnancy
* Any implanted electrical device
* Any significant dermatological/infectious condition of the ear

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thangam Venkatesan, Principal Investigator — MCW
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
NA. Our data will only be made available to the study team at the Medical College of Wisconsin as noted in the IRB

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Placebo Group
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Placebo Group | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (7) | 34.5 (2.1) | 32.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Abdominal Pain
Description: Abdominal pain will be assessed through Visual Analog Scale with the score of ranging from 0 to 10, with 0 being the least and 10 being the worst pain.
Time Frame: The change in abdominal pain will be measured at baseline (before intervention) and then at 2 hours, 24 hours and at 5 days post intervention.
Population: Data was not collected due to entry problem with participants not adding identifying information with their logs.
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Need for Opioids Between Device and Sham
Description: The amount of opioids used by the patient will be recorded in all subjects and will be converted into morphine equivalents for comparison
Time Frame: The dose of opioids use ( morphine equivalent) will be measured at baseline (before intervention) and then at 2 hours, 24 hours and at 5 days post intervention.
Population: Data not collected.
Groups:
- Sham Group: The sham was similar to the intervention device in all respects except that there was no current delivered.
Arm/Group | Intervention Group | Sham Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Index for Nausea, Vomiting and Retching (INVR) Scores
Description: The severity of daily nausea, vomiting and retching will be assessed using the Index for Nausea, Vomiting and Retching (INVR). This is a validated tool to measure the severity of nausea, vomiting and retching. The scores range from 0-32 with 0 being the least severe and 32 being the most severe.
Time Frame: The INVR scores will be assessed be measured at baseline (before intervention) and then at 2 hours, 24 hours and at 5 days post intervention.
Reporting Status: Not Posted

4. Secondary Outcome: Length of Stay in the Hospital (LOS)
Description: Hospital Length of stay (LOS) in days which refers to the no of days that the patient was admitted in the inpatient ward or unit
Time Frame: LOS will be determined at end of 1 month
Reporting Status: Not Posted

5. Secondary Outcome: Patient Satisfaction
Description: A validated patient satisfaction score will be used
Time Frame: Patient satisfaction will be assessed at end of 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: This was done for 6 months
Description: This study was performed in the emergency department/hospital setting and hence a hospitalization or emergency department visit would not qualify as an adverse event in this study.
Groups:
- Sham Group: The Sham device is a non-invasive percutaneous electrical nerve field stimulation (PENFS) applied to the external ear. It is similar to the sham but does not deliver any electrical stimulation.
  This is placed on the ear as per standard protocol at the beginning of the study and removed by the patient after 5 days.
Arm/Group | Intervention Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated due to COVID. There was a multidisciplinary team that was assembled which consisted of the emergency departments, hospitalists and gastroenterologist. Due to the unprecedented crisis which involved lockdowns, and furloughs we lost our resources and the ability to continue the study or collect data.

We will be revising our plan on lessons learned during this study and will start a new protocol with changes and to solve COVID-related issues that are a barrier.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT04721171/Prot_SAP_000.pdf